CLINICAL TRIAL: NCT00295568
Title: Contribution of Interhemispheric Inhibition to Motor Learning
Brief Title: Interaction of Right and Left Brain Hemispheres in Learning Precision Hand Movements
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060095; 06-N-0095
Record Dates: First submitted 2006-02-23; First posted 2006-02-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-12

CONDITIONS: Interhemispheric Inhibition
Keywords: Transcranial Magnetic Stimulation (TMS); Motor Learning; Accuracy; Tracking Motor Task; Healthy Volunteer; HV

SUMMARY:
This study will examine how the two sides of the brain interact when learning precision hand movements. Both sides of the brain are active when a person performs an accurate hand movement. This study will look at the extent to which the two brain hemispheres interact when learning accurate hand movements.

Healthy, right-handed normal volunteers 18 - 40 years of age may be eligible for this study. Candidates are screened with a clinical and neurological examination.

Participants are randomly assigned to one of two groups - precision or non-precision hand movements. All participants undergo the following procedures:

* Force precision task: Subjects are press a small device between the thumb and index finger. The force produced with the fingertips is translated onto a computer screen. Subjects track a white line passing on the screen with their fingertips.
* Paired-pulse transcranial magnetic stimulation (TMS): A wire coil is held to the subject's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil. The effect of paired-pulse TMS on the muscles is detected with electrodes taped to the skin on the arms or legs.
* Surface electromyography (EMG): This test measures the electrical activity of muscles. For this test, electrodes are filled with a gel and taped to the skin over the muscle to be tested.

The study involves six sessions. Sessions 1-5 are on consecutive days; session 6 is one week after session 5.

* Session 1: Familiarization with the motor task and baseline measurements, including error rate, EMG, and paired-pulse TMS
* Session 2: Training in the motor task and repeat measurements as in session 1
* Session 3: Training and measurements as in session 2
* Session 4: Training and measurements as in session 2
* Session 5: Training and measurements as in session 2
* Session 6: Measurements only

DETAILED DESCRIPTION:
The purpose of this protocol is to investigate the changes in interhemispheric inhibition (IHI) between human motor cortices with learning of performance of an accurate motor task (pinch force control). Performing a simple motor task is associated with activation in the contralateral motor areas. Activation of the ipsilateral motor/premotor cortex might be elicited by performing more challenging and difficult unimanual motor tasks. However, the functional role played by this ipsilateral activation has been controversial, and is felt to be more prominent with more complex tasks. Several studies using paired-pulse transcranial magnetic stimulation (TMS) revealed a significant IHI from the active upon the non-active hemisphere. Together these results suggested IHI between motor cortical areas may play a critical role in motor control and could influence manual dexterity. Taking these into account, it raises the interesting question of whether the IHI balance between both motor cortices is progressively modified during the learning phase of an accurate motor task. We hypothesize that learning to perform a tracking motor task requiring accurate control of pinch force generation (Tracking accurate), will increase IHI from the "learning" to the "non-learning" hemisphere to a larger extent than learning to perform a less precise tracking motor task (Tracking non-accurate). The primary outcome measure will be the amount of changes in IHI from the "learning" to the "non-learning" hemisphere as a function of learning both motor tasks.

ELIGIBILITY:
* INCLUSION CRITERIA

Healthy volunteers will be eligible for the study if they are:

* are between the ages of 18-40 years;
* are right-handed;
* are able to perform tasks required by the study;
* are willing and able to give consent

EXCLUSION CRITERIA

Healthy volunteers will not be eligible for the study if they:

* are unable to perform the tasks;
* are left-handed;
* have a history of neurological and psychiatric illness, or of alcohol or drug abuse or severe language disturbances or serious cognitive deficits;
* have uncontrolled medical problems, such as heart, lung or kidney disease, epilepsy or diabetes mellitus, have severe tactile deficits (defined by Frey filaments exerting a force of 4 N to the distal pad of the finger);
* have a cardiac pacemaker, intracardiac lines, implanted medication pumps, neural stimulators, metal in the cranium, with the exception of dental braces.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46
Dates: Start 2006-02-17; Study Completion 2009-01-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kim SG, Ashe J, Hendrich K, Ellermann JM, Merkle H, Ugurbil K, Georgopoulos AP. Functional magnetic resonance imaging of motor cortex: hemispheric asymmetry and handedness. Science. 1993 Jul 30;261(5121):615-7. doi: 10.1126/science.8342027.
- [Background] Beltramello A, Cerini R, Puppini G, El-Dalati G, Viola S, Martone E, Cordopatri D, Manfredi M, Aglioti S, Tassinari G. Motor representation of the hand in the human cortex: an f-MRI study with a conventional 1.5 T clinical unit. Ital J Neurol Sci. 1998 Oct;19(5):277-84. doi: 10.1007/BF00713853. PMID 10933447
- [Background] Roland PE, Skinhoj E, Lassen NA, Larsen B. Different cortical areas in man in organization of voluntary movements in extrapersonal space. J Neurophysiol. 1980 Jan;43(1):137-50. doi: 10.1152/jn.1980.43.1.137. PMID 7351548